CLINICAL TRIAL: NCT06039449
Title: A Study to Evaluate the Efficacy and Safety of VYD222 for Prevention of COVID-19 (CANOPY)
Brief Title: A Study to Investigate the Prevention of COVID-19 WithVYD222 in Adults with Immune Compromise and in Participants Aged 12 Years or Older Who Are At Risk of Exposure to SARS-CoV-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Invivyd, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VYD222-PREV-001
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: COVID-19; SARS-CoV-2
Keywords: Immune Compromise; VYD222; SARS-CoV-2 Monoclonal Antibody; COVID-19 Prevention
MeSH Terms: conditions — COVID-19 | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only applies to Cohort B
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort A VYD222 (Experimental)
  Interventions: Drug: VYD222 (pemivibart)
- Cohort B VYD222 (Experimental)
  Interventions: Drug: VYD222 (pemivibart)
- Cohort B Placebo (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: VYD222 (pemivibart) — Participants will be dosed on Day 1 followed by redosing at Month 3 (approximately 90 days) with VYD222.
  Arms: Cohort A VYD222; Cohort B VYD222
Drug: Normal saline — Participants will be dosed on Day 1 followed by redosing at Month 3 (approximately 90 days) with Placebo.
  Arms: Cohort B Placebo

SUMMARY:
A study to investigate the prevention of COVID-19 with VYD222 in adults with immune compromise and in participants aged 12 years or older who are at risk of exposure to SARS-CoV-2

ELIGIBILITY:
Inclusion Criteria:

* Is an adult aged ≥18 years or an adolescent aged 12 to <18 years and weighs at least 40 kg at the time of Screening.
* Tests negative for current SARS-CoV-2 infection by local antigen test or RT-PCR at the time of Screening.
* For Cohort A, has significant immune compromise from causes including solid tumor or hematologic malignancies, chimeric antigen receptor (CAR)-T-cell therapy or hematopoietic stem cell transplant, primary immunodeficiency, advanced HIV infection, or receiving qualifying immunosuppressive therapies.
* For Cohort B, is at risk of acquiring SARS-CoV-2 due to regular unmasked face-to-face interactions in indoor settings.
* Agrees to defer receipt of any COVID-19 vaccination or booster for a minimum of 28 days after dosing.
* Note: unless specified by Cohort, the criteria apply to both Cohorts

Exclusion Criteria:

* For Cohort B: Prior receipt of a COVID-19 vaccine or booster within 120 days before randomization.
* Prior receipt of convalescent plasma or a mAb to SARS-CoV-2 active against currently circulating variants, including in the setting of a clinical trial, within 120 days before randomization.
* Prior known or suspected SARS-CoV-2 infection within 120 days before randomization.
* Exposure to someone with known or suspected SARS-CoV-2 infection in the 5 days before randomization.
* Is acutely ill or has any symptoms suggestive of infection, in the opinion of the Investigator.

Note 1: Other protocol defined inclusion/exclusion criteria apply Note 2: Unless specified by Cohort, the criteria apply to both Cohorts

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Cohort A - Incidence of treatment emergent adverse events | Through Month 12
Cohort A - Ratio of SARS-CoV-2 sVNA titer against a relevant variant following VYD222 administration at Day 28 compared to a prespecified SARS-CoV-2 sVNA titer threshold. | Day 28
Cohort B - Incidence of treatment emergent adverse events | Through Month 12

SECONDARY OUTCOMES:
Cohort A - Proportion of participants with sVNA titer against a relevant variant following VYD222 administration at Day 28 above a prespecified SARS-CoV-2 sVNA titer threshold. | Day 28
Cohort A - sVNA titer by timepoint following VYD222 administration | Through Month 12
Cohort A - Proportion of participants with sVNA titer against a relevant variant following VYD222 administration above a minimum SARS-CoV-2 sVNA threshold by timepoint | Through Month 12
  The minimum SARS-CoV-2 sVNA titer threshold will be prespecified prior to analysis.
Cohort A - ADAs against VYD222 | Through Month 12
Cohort A - Serum concentrations (PK) of VYD222 | Through Month 12
Cohort A - Proportion of participants with RT-PCR-confirmed symptomatic COVID-19 | Through Month 12
  RT-PCR-confirmed symptomatic COVID-19 is defined as RT-PCR-confirmed SARS-CoV-2 with an onset of symptoms occurring no more than 14 days from the date of the positive RT-PCR test sample collection, COVID-19-related hospitalization, or all-cause death.
Cohort B - Ratio of SARS-CoV-2 sVNA titer against a relevant variant following VYD222 administration at Day 28 compared to a prespecified SARS-CoV-2 sVNA titer threshold. | Day 28
Cohort B - Proportion of participants with sVNA titer against a relevant variant following VYD222 administration at Day 28 above a prespecified SARS-CoV-2 sVNA titer threshold. | Day 28
Cohort B - sVNA titer by timepoint following VYD222 administration | Through Month 12
Cohort B - Proportion of participants with sVNA titer against a relevant variant following VYD222 administration above a minimum SARS-CoV-2 sVNA threshold by timepoint | Through Month 12
  The minimum SARS-CoV-2 sVNA titer threshold will be prespecified prior to analysis.
Cohort B - COVID-19-related hospitalization or COVID-19-related death within 28 days of symptom onset | Through Month 12
Cohort B - COVID-19-related death | Through Month 12
Cohort B - Serum concentrations (PK) of VYD222 | Through Month 12
Cohort B - ADAs against VYD222 | Through Month 12

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - INVIVYD Investigative Site, Fullerton, California
  - INVIVYD Investigative Site, Long Beach, California
  - INVIVYD Investigative Site, Rolling Hills Estates, California
  - INVIVYD Investigative Site, San Diego, California
  - INVIVYD Investigative Site, Clearwater, Florida
  - INVIVYD Investigative Site, Miami, Florida
  - INVIVYD Investigative Site, St. Petersburg, Florida
  - INVIVYD Investigative Site, Atlanta, Georgia
  - INVIVYD Investigative Site, Hinesville, Georgia
  - INVIVYD Investigative Site, Oak Brook, Illinois
  - INVIVYD Investigative Site, Silver Spring, Maryland
  - INVIVYD Investigative Site, Burlington, Massachusetts
  - INVIVYD Investigative Site, Morrisville, North Carolina
  - INVIVYD Investigative Site, Salisbury, North Carolina
  - INVIVYD Investigative Site, Edmond, Oklahoma
  - INVIVYD Investigative Site, Yukon, Oklahoma
  - INVIVYD Investigative Site, Beaumont, Texas
  - INVIVYD Investigative Site, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolfe CR, Cohen J, Mahoney K, Holmes A, Betancourt N, Gupta D, Tosh K, Narayan K, Campanaro E, Katz C, Phelan AM, Yalcin I, Wingertzahn M, Hawn P, Schmidt P, Li Y, Popejoy M. Safety and Efficacy of Pemivibart, a Long-Acting Monoclonal Antibody, for Prevention of Symptomatic COVID-19: Interim Results From a Phase 3 Randomized Clinical Trial (CANOPY). Clin Infect Dis. 2025 Oct 6;81(3):439-450. doi: 10.1093/cid/ciaf265. PMID 40410927